CLINICAL TRIAL: NCT06167889
Title: Gender-specific Impact Factors on Elderly Disability and Cognitive Impairment: A Retrospective Cohort Study
Brief Title: A Study of Gender-specific Impact Factors on Elderly Disability and Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Fang Tang (Other)
Responsible Party: Sponsor-Investigator, Fang Tang, Doctor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(140)
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Aging
Keywords: Elderly; Disability; Cognitive impairment; Gender-specific
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort based on Shandong Provincial Qianfoshan Hospital Healthcare Big Data Platform: A retrospective cohort based on Shandong Provincial Qianfoshan Hospital Healthcare Big Data Platform is conducted to collect data and to explore the gender differences and influencing factors of disability and cognitive impairment among the elderly.
- Retrospective cohort from CLHLS: The data from the China Longitudinal Healthy Longevity Survey (CLHLS) was used to further validate the results.

SUMMARY:
Elderly disability and cognitive impairment rates were different between elderly man and woman. Sex-specific risk factors and observed gender differences across the lifespan were associated with different degrees of cognitive and activity of daily living function decline between men and women. However, some of these viewpoint remains controversial.

The aim of this study is to explore the gender differences and influencing factors of disability and cognitive impairment among the elderly.

DETAILED DESCRIPTION:
With the rapid increase in the aging population in China, age-related cognitive impairment and disability has become a pressing public health concern. A number of large-scale studies in China and abroad have shown that the average life expectancy of women elderly is higher than men, but the rates of disability and cognitive impairment are higher. However, it is lack of exploration of the factors associated with the gender-specific of disability and cognitive impairment.

The aim of this study is to explore the gender differences and influencing factors of disability and cognitive impairment among the elderly. A retrospective cohort based on Shandong Provincial Qianfoshan Hospital Healthcare Big Data Platform is conducted to collect data. And the data from the China Longitudinal Healthy Longevity Survey (CLHLS) was used to further validate the results.

ELIGIBILITY:
Inclusion Criteria:

1.The elderly aged 65 and above.

Exclusion Criteria:

1. Lack of diagnostic information.
2. Missing key influencing factors such as gender and age.
3. Hearing or linguistic impairment.
4. Comatose patients.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The elderly aged 65 and above in the China Longitudinal Healthy Longevity Survey (CLHLS) database and the elderly with health care neurology visits recorded in Shandong Provincial Qianfoshan Hospital Healthcare Big Data Platform
Sampling Method: Non-Probability Sample
Enrollment: 23640 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Disability | 2002-2023
  We identified disability according to the Katz index. This Katz index includes six activities of daily life: bathing, transferring, dressing, eating, toileting, and continence. Disability was defined as needing help with at least one of the six activities of daily life.
Cognitive impairment | 2002-2023
  The main outcome was assessed by the Chinese version of the Mini-Mental State Examination (CMMSE).For participants who had never received education, an MMSE score of 17 or less was considered as cognitive impairment; for those who had less than 6 years of education, an MMSE score of 20 or less was considered as cognitive impairment; and for those who had more than 6 years of education, an MMSE score of 24 or less was considered as cognitive impairment. For each level of education, scores above the threshold were considered cognitively normal.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Tang, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China